CLINICAL TRIAL: NCT02416362
Title: Immediate Effects of Whole Body Vibration on Neuromuscular Performance of Quadriceps Femoris and Balance of Healthy Women: a Randomized Controlled Trial
Brief Title: Immediate Effects of Whole Body Vibration on Neuromuscular Performance of Quadriceps Femoris and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Associeted Professor and Researcher, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DTB2014
Record Dates: First submitted 2015-03-17; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Neuromuscular Performance and Balance
Keywords: Postural Balance; Electromyography; Torque

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The control group (No vibration) will hold an exercise protocol on the vibration platform, which is to stay on one foot on the non-dominant leg, with the knee held in 40 ° of flexion, hands together to the body and the trunk in the erect position. Altogether, the participant will perform 11 sets of 30 seconds with a rest interval of 30 seconds between sets. The knee angle will be monitored throughout the protocol by the second reviewer with a goniometer so that there is no change in it. The vibrating platform will remain off throughout intervention.
- GE1 (Experimental): The GE1 (Vibration at 30 Hz) group will hold an exercise protocol on the vibration platform, which is to stay on one foot on the non-dominant leg, with the knee held in 40 ° of flexion, hands together to the body and the trunk in the erect position. Altogether, the participant will perform 11 sets of 30 seconds with a rest interval of 30 seconds between sets. The knee angle will be monitored throughout the protocol by the second reviewer with a goniometer so that there is no change in it. During the sets the vibrating platform will be turned on at a vibration frequency of 30 Hz.
  Interventions: Other: Vibration at 30 Hz
- GE2 (Experimental): The GE1 (Vibration at 50 Hz) group will hold an exercise protocol on the vibration platform, which is to stay on one foot on the non-dominant leg, with the knee held in 40 ° of flexion, hands together to the body and the trunk in the erect position. Altogether, the participant will perform 11 sets of 30 seconds with a rest interval of 30 seconds between sets. The knee angle will be monitored throughout the protocol by the second reviewer with a goniometer so that there is no change in it. During the sets the vibrating platform will be turned on at a vibration frequency of 50 Hz.
  Interventions: Other: Vibration at 50 Hz

INTERVENTIONS:
Other: Vibration at 30 Hz — During the exercise protocol, the vibration platform will be turned on at a vibration frequency of 30 Hz.
  Arms: GE1
Other: Vibration at 50 Hz — During the exercise protocol, the vibration platform will be turned on at a vibration frequency of 50 Hz.
  Arms: GE2

SUMMARY:
The purpose of this study is to analyze the immediate effects of two exercise protocols on the vibration platform, on the strength of the thigh muscles, joint position sense of the knee and balance in healthy subjects.

DETAILED DESCRIPTION:
Design and research site: This is a randomized and blinded clinical trial held at the Laboratory of Neuromuscular Performance of the Department of Physical Therapy, Federal University of Rio Grande do Norte (UFRN). Characterization of the sample: The sample consisted of 60 women randomly divided into 3 distinct groups. Ethical aspects: For its implementation, this project was submitted to the Research Ethics Committee (REC) of the Federal University of Rio Grande do Norte. Was respected and ensured the autonomy and anonymity of participants, as well as your privacy as confidential data, as governed Resolution 196/96 of the National Health Council and the Helsinki declaration for human research. Instruments: Stationary bicycle (Ergo-Fit, ErgoCycle 167, Pirmasens, Germany); computerized baropodometry platform Eclipse 3000 model (Guy-Capron® SA, France); vibrating platform model Power Plate® pro5 ™; signal conditioning module (Telemyo direct transmission system) 8-channel (Noraxon, USA); self-adhesive electrode active surface (Noraxon, USA); isokinetic dynamometer (Biodex Multi-Joint System 4, Biomedical Biodex System Inc.®, New York, USA). Procedures: There was a previous pilot study for adequacy of any research procedures and the training of evaluators. The volunteers were informed about the procedures to be performed in the research, signed the informed consent form, fill in an evaluation form with anthropometric data and personal examination of members. Evaluations were performed before and after the intervention protocol. Initially, all the volunteers executed a warming exercise on a stationary bike for 5 minutes. Postural balance: the volunteers were placed standing on the baropodometry platform, supported in the non-dominant member and with the knee kept at 20 ° of flexion. The dominant member remained with the knee in 90 ° of flexion. The evaluation was repeated 3 times, being considered for analysis the average of the two best measures. The evaluation time was 20 seconds on an acquisition frequency of 20 Hz with a period of 1 minute break between tests. Previously the participant was allowed to become familiar with the equipment. Joint position sense: the volunteer was positioned sitting on the dynamometer, stabilized by braces and with the device axis aligned with the knee evaluated. The apparatus of the lever arm was attached to the distal leg. Then, the volunteer was instructed to perform a knee extension member starting with 90 ° of flexion. When the 45 target angle wass reached, the dynamometer arm remained in this position, keeping it for 5 seconds, so that the voluntary noticed which the angle to be achieved. Finally, prompted an active extension from 90 ° knee flexion (1 / s) to the target angle, the second trial of the subject. At that moment, the volunteer should trigger a device to record the angle reached. Torque rating: keeping the same previous position, the normalization of the electromyographic signal was held, where the subject performed two maximal voluntary isometric contractions of knee extension at an angle of 60 ° for 5s, with one-minute interval between each repetition. Then the concentric evaluation was conducted, with 5 maximal contractions for knee flexion and extension at 60 ° / s, starting from 90 ° flexion up to full extension. Electromyographic activity: emg was collected concurrently with exercise protocols on the platform, as well as during the torque rating. The volunteers were submitted for shaving and cleaning the skin with 70% alcohol before attaching the electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Healthy
* Engaging in physical activity involving lower limbs at least 3 times per week
* Exhibiting ankle, hip and knee joint integrity of the non-dominant limb
* No history of muscle or joint injuries in the assessed limb in the last 6 months, or neurological, visual and/or non-corrected auditory impairments

Exclusion Criteria:

* Auto-desistance
* Referring pain or discomfort during the procedures for collection
* Not perform assessment procedures correctly in order to make it impossible to capture the data.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Muscle Performance measured through isokinetic dynamometry | Baseline, immediately after the intervention protocol
  The muscle performance will be measured through isokinetic dynamometry and the variables analyzed will be peak torque normalized for body weight, mean power, total work and time to peak torque.

SECONDARY OUTCOMES:
Proprioception measured through joint position sense in the isokinetic dynamometer | Baseline, immediately after the intervention protocol
  The proprioception will be measured through joint position sense
Muscle activation measured through surface electromyography | Baseline, immediately after the intervention protocol
  Measured by surface electromyography
Balance measured through baropodometry | Baseline, immediately after the intervention protocol
  Measured by baropodometry

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] Borges DT, Macedo LB, Lins CA, Brasileiro JS. Immediate effects of whole-body vibration on neuromuscular performance of quadriceps and oscillation of the center of pressure: A randomized controlled trial. Man Ther. 2016 Sep;25:62-8. doi: 10.1016/j.math.2016.06.005. Epub 2016 Jun 16. PMID 27422599